CLINICAL TRIAL: NCT05108454
Title: Evaluation of a Business Model of Multiple Micronutrient Supplementations (MMS) Project for Bangladeshi Pregnant Women
Brief Title: Multiple Micronutrient Supplementation (MMS) Evaluation Among Bangladeshi Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Children's Investment Fund Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PR-21001
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Infant, Low Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Pregnant women who received MMS from the SMC program
  Interventions: Drug: Multiple micronutrient supplementation
- Comparison: Pregnant women who did not receive MMS

INTERVENTIONS:
Drug: Multiple micronutrient supplementation — Multiple Micronutrient Supplements (MMS) is a nutritional supplement for use during pregnancy based on United Nations International Multiple Micronutrient Antenatal Preparation (UNIMMAP) formulation following WHO specification. It contains 15 micronutrients including Iron and Folic Acid (IFA) at dosages that approximate the recommended dietary allowances for pregnancy.
  Other Names: MMS
  Groups: Intervention group

SUMMARY:
Maternal nutrition profoundly affects foetal growth, development, and subsequent infant birth weight. Babies with low birth weight (LBW) have an elevated risk of death in infancy and later childhood. A recent systematic review revealed that multiple micronutrient supplementations (MMS) could reduce the risk of LBW by 13% in comparison with iron and folic acid (IFA). Based on this newer evidence, the World Health Organization (WHO) recommended MMS during a pregnancy instead of IFA, with consideration of the country context-specific research. However, little progress is being achieved in ensuring adequate MMS coverage to improve pregnancy outcomes. Based on the WHO recommendation, CIFF awarded the Social Marketing Company (SMC) to set up a sustainable business model with affordable and quality MMS to pregnant women in Bangladesh over a period of 5 years through SMC's pharmacy networks. The investigators propose to develop an evaluation design including both process and outcome evaluation to evaluate the implementation and effect of the MMS by the SMC in Bangladesh. The evaluation study will comprise both process and outcome evaluation, complementing each other. The design will be a quasi-experimental cluster-based open cohort, two-arm, mixed-methods design. The evaluation would take place in 5 divisions of Bangladesh.

DETAILED DESCRIPTION:
Background: a. Burden: Maternal nutrition profoundly affects foetal growth, development, and subsequent infant birth weight. Babies with low birth weight (LBW) have an elevated risk of death in infancy. Furthermore, these babies have a higher risk of stunting or linear growth failure and slower mental development in childhood. b. Knowledge gap: A recent systematic review revealed that multiple micronutrient supplementations (MMS) could reduce the risk of LBW by 13% in comparison with iron and folic acid (IFA). Based on this newer evidence, the World Health Organization (WHO) has updated the antenatal nutrition recommendations. Now, MMS is recommended during a pregnancy instead of IFA, with consideration of the country context-specific research. However, little progress is being achieved in ensuring adequate MMS coverage to improve pregnancy outcomes. Furthermore, the MMS tablets are expensive compared to the IFA, which might hinder the uptake of the MMS by the people. c. Relevance: Based on the WHO recommendation, CIFF awarded the Social Marketing Company (SMC) to set up a sustainable business model with affordable and quality MMS to pregnant women in Bangladesh over a period of 5 years through SMC's pharmacy networks. The investigators propose to develop an evaluation design including both process and outcome evaluation to evaluate the implementation and effect of the MMS by the SMC in Bangladesh.

Hypothesis: The prevalence of LBW will be reduced by 5% point in the intervention group compared to the control group by the end of the 5-year program.

Objectives: Outcome evaluation- To evaluate the effectiveness of market-based distribution of MMS intervention on the prevalence of low birth weight (less than 2500 g) in the infants born to women in the intervention area who received the intervention compared to control areas Process evaluation- To measure the fidelity, reach and mechanism of impact of the intervention

Methods: The evaluation study will comprise both process and outcome evaluation, complementing each other. The design will be a quasi-experimental cluster-based open cohort, two-arm, mixed-methods design. The evaluation would take place in 5 divisions of Bangladesh: Barishal, Chattogram, Dhaka, Rajshahi, and Sylhet. For outcome evaluation: Eligible pregnant women will be approached for recruitment with proper consent. Right after recruitment, a baseline data collection will be conducted using a structured questionnaire along with anthropometric measurements. The recruited participants will be followed up until the end of their pregnancy. After successful delivery of a baby, an endpoint data collection will be done along with birth weight measurement of the baby. Data from the control areas will be collected following the same guideline to maintain consistency. The process evaluation will be carried out concurrently to monitor the program activities. This will follow a mixed-method design, including both quantitative and qualitative components. The participants will be recruited from the same area where activity for outcome evaluation will be ongoing. The investigators will focus on the fundamental aspects of process evaluation that includes- (a) understanding the health promotion program and how it is supposed to work, (b) defining the purposes for the process evaluation, and (c) considering program characteristics and context and how these may affect implementation.

Outcome measures/variables: The key variable for outcome evaluation is the measurement of birth weight. Key variables for process evaluation are fidelity, reach, and mechanism of impact of the intervention (MMS).

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy identified/reported through ultrasonogram during ANC or other available medical proof
* Absence of severe malnourishment/known chronic diseases- respiratory illness, hypertension, diabetes, TB, haemoglobinopathy, etc. through self-reporting and available documents
* Participant willingness to participate
* Provide at least two mobile numbers to contact
* The place of delivery has been decided

Exclusion Criteria:

* Non-pregnant
* Declined to participate

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women.
Study Population: Pregnant mothers live in either intervention or control areas in any trimester of pregnancy.
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Low birth weight babies | November 2021 to June 2024
  Babies born with birth weight less than 2500 grams

SECONDARY OUTCOMES:
Percentage of Preterm children | November 2021 to June 2024
  Babies born less than 37 weeks of gestation
Number of pregnant women with MMS side effects, compliance, & adverse perinatal outcomes | November 2021 to June 2024
  MMS side effects: Any side effects of MMS reported by the pregnant mothers. MMS compliance: Pregnant mothers intake of 180 MMS tablets once a day for 6 months.
  Adverse perinatal outcomes: Any maternal and child health complication before and after child delivery.
Percentages of contact and effective coverage for the intervention group | November 2021 to June 2024
  Reach and utilization of MMS and compliance of pregnant women who consumed MMS
Number of pregnant women with their duration of gestation | November 2021 to June 2024
  Duration of pregnancy in months among the pregnant women at both intervention and control group

CONTACTS AND LOCATIONS:
Overall Officials: Muttaquina Hossain, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
We will strictly follow the icddr,b's ethical guideline and practice to ensure the confidentiality of information collected through this study. The name and phone number(s) of the respondent will not be included in the data set. All data will be stored in a password-protected PC having access to only selected individual(s) using STATA software in a specified drive. After a specific time, data be backed up in three places such as another drive in the same computer, in a PI's computer, and in an additional hard drive which will be placed in a secured location. The information collected from this study may be shared with other researchers if needed only for research purposes, however, it will be strictly followed to maintain confidentiality and privacy and as per the icddr,b's data access policy.
Supporting Information: Study Protocol, SAP
Time Frame: After the study completes.
Access Criteria: icddr,b study investigators.

REFERENCES:
- [Derived] Hossain M, Sanin KI, Haque MA, Mbuya MNN, Ghosh S, Aksari S, Gibson S, Neufeld L, Bipul M, Matubbar S, Rahman MM, Khondker R, Salasibew M, Ahmed T. Evaluating the impact of a countrywide, market-based roll-out of multiple micronutrient supplementation on low birth weight in Bangladesh: protocol for a two-arm, quasi-experimental and mixed-methods evaluation study. BMJ Open. 2022 May 30;12(5):e060230. doi: 10.1136/bmjopen-2021-060230. PMID 35636782